CLINICAL TRIAL: NCT03368898
Title: Comparison of Estradiol Valerate (E2V), Levonorgestrel- Intrauterine Device (LNG-IUD) and Oral Micronized Progesterone Therapy on Health-related Quality of Life in Premenopausal Women With Heavy Menstrual Bleeding
Brief Title: Quality of Life in Premenopausal Women With Heavy Menstrual Bleeding
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Ismail Alay, principal investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: HMBSYMPTOM
Record Dates: First submitted 2017-11-29; First posted 2017-12-11 (Actual); Results first posted 2020-09-03 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Heavy Menstrual Bleeding
MeSH Terms: conditions — Menorrhagia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Estradiol valerate: Women who were treated with E2V for HMB for 3 months.
- LNG-IUD: Women who were treated with LNG-IUD for HMB for 4 years.
- Micronized Progesterone: Women who were treated with Micronized Progesterone for HMB for 3 months.

SUMMARY:
Heavy menstrual bleeding or menorrhagia, is a common problem on women's lives and can burden both patients and health care systems. HMB is defined as cyclic heavy vaginal bleeding. Hormonal treatment of heavy menstrual bleeding (HMB) is also endorsed as the first line treatment in several international guidelines. The effects of these therapies on bleeding related quality of life are not well known. The aim of the present study is compare the effect of Estradiol Valerate/Dienogest (E2V/DNG), Levonorgestrel-Intrauterine Device (LNG-IUD) and oral micronized progesterone treatment on bleeding pattern, cycle control, menopausal symptoms and patient satisfaction of women with HMB.

DETAILED DESCRIPTION:
Women who were admitted and treated for HMB were asked to participate in this comparative study. Women were eligible for entry if they had self-described heavy menstrual bleeding, had a regular cycle, had completed their family and were 40-50 years old at initial assessment.

After a thorough physical examination and ultrasonographic evaluation, all women underwent endometrial biopsy before the study by using a Pipelle endometrial suction curette to rule out any organic endometrial pathology. Blood samples were analysed to test for hemoglobin (Hb), hematocrit (Hct), ferritin, serum iron and iron-binding capacity and coagulation tests such as prothrombin time and activated partial thromboplastin time.

The study was approved by the Institutional Review Board and Local Ethics Committee. After they gave written informed consent, patients who fulfilled eligibility criteria were recruited to one of the following 3 groups:

Group 1: Women who were treated with estradiol valerate/dienogest regimen for heavy menstrual bleeding. 28 days of E2V/DNG was administered using a dynamic dosing regimen. (E2V 3 mg on days 1-2, E2V 2 mg/DNG 2 mg on days 3-7, E2V 2 mg/DNG 3 mg on days 8-24, E2V 1 mg on days 25-26 and placebo on days 27-28).

Group 2: Women who were treated with LNG-IUD for heavy menstrual bleeding. LNG-IUD is containing 52 mg levonorgestrel at initial placement and releases 20 microgram levonorgestrel per day. This is approved for 5 years of use by the US FDA for treatment of HMB.

Group 3: Women who were treated with oral Micronized Progesterone 200 mg for heavy menstrual bleeding. Cyclic, luteal-phase administration of progestin remained a widely used but little research treatment strategy for HMB for several decades.

None of the recruited patients were not prescribed oral iron preparations and patients who were symptomatic because of anemia (hb<10 mg/dl) were excluded.

Baseline characteristics of women are age (years), body mass index, parity, current smoker, days of bleeding, length of cycle (days), number of days of heavy bleeding, number of days of painful bleeding, unable to leave house on heaviest days, number of days housebound, number of nights disturbed, Pictorial Bleeding Assessment Chart (PBAC) score (A monthly score of 100 or more on this chart is significantly associated with heavy menstrual bleeding of more than 80 ml per cycle, as measured by the alkaline haematin method), endometrial thickness at time of treatment (mm), uterine size (length x width).

The Exclusion criteria are

1. ultrasound abnormalities (submucosal fibroids, intramural fibroids greater than 3 cm in diameter, large subserosal fibroids, endometrial polyps);
2. laboratory abnormalities (follicle stimulating hormone level higher than 40 iu/l, adverse endometrial histology)
3. hysteroscopic abnormalities (submucosal fibroids, endometrial polyps),
4. incidental adnexal abnormality on ultrasound,
5. severe intermenstrual bleeding, severe dysmenorrhoea, severe premenstrual pain, chronic pelvic pain,
6. medical contraindications to either study treatment,
7. previous endometrial ablation or resection,
8. uninvestigated postcoital bleeding
9. untreated abnormal cervical cytology.
10. pregnancy; lactation; occurrence of <3 menstrual cycles following childbirth, abortion or lactation;
11. current use of an intrauterine device; hypersensitivity to any of the study drug ingredients and known or suspected malignant or premalignant disease.
12. systemic diseases like hypertension, diabetes, thyroid diseases or coronary artery diseases; and history of previous medication for menorrhagia
13. using anticoagulant drugs

Women who were recruited the study will be assessed at 1,3 and 6 months with Hot Flush Rating Scale (HFRS), Menopause Rating Scale (MRS), menorrhagia multi-attribute scale (MM-AS), pictorial bleeding assessment chart and blood sample analysis.

The primary outcomes assessed

1. Hot flush rating scale: Measures included the HFRS, a self-report measure of frequency and problem rating of Hot Flushes/Night Sweats over the past week. Problem rating is calculated as the mean of the scores on three ten-point scales assessing the extent to which Hot Flushes/Night Sweats are problematic, distressing and causing interference in daily life. Scores for the problem rating range between 1 and 10, with higher scores indicating more problematic Hot Flushes/Night Sweats. The HFRS has been found to have reasonable test-retest reliability and good concurrent validity.
2. Menopause rating scale: The Menopause Rating Scale (MRS) is a questionnaire that assesses the presence and intensity of 11 menopausal symptoms. These are grouped into three subscales: the somatic subscale: assessing hot flushes/sweating, heart discomfort, sleeping problems, and muscle and joint discomfort (items 1-3 and 4 respectively); the psychological subscale: assessing depressive mood, irritability, anxiety, and physical and mental exhaustion (items 4-7 respectively); and the urogenital subscale: assessing sexual problems, bladder problems and vaginal dryness (items 8- 10, respectively). Each of the 11 items can be rated by the participant from 0 (not present) to 4 (1 ¼ mild, 2 ¼ moderate, 3 ¼ severe and 4 ¼ very severe). The scores obtained for each individual item are summed to provide the corresponding total subscale score. The sum of subscales scores provide the total MRS score. Higher scores are indicative of more severe symptoms. Indeed values above 8 (somatic), 6 (psychological), 3 (urogenital) and 16 (total MRS) were defined as severe.

The secondary outcomes assessed

1. Quality of life as measured by menorrhagia multi-attribute scale: which is designed to measure the effect of menorrhagia on six domains of daily life (practical difficulties, social life, psychological health, physical health, work and daily routine, and family life and relationships). Summary scores, which range from 0 (severely affected) to 100 (not affected)
2. Menstruation, by pictorial bleeding assessment chart
3. Haemoglobin levels were also measured at pre-treatment,1, 3 and 6 months.
4. Adverse event (Breast pain, Headache, Acne, Alopecia, Migraine, Increase in body weight…)

ELIGIBILITY:
Inclusion Criteria:

* women who self described heavy menstrual bleeding
* women who completed their family
* have cyclic menstruation
* 40 to 50 years old

Exclusion Criteria:

1. ultrasound abnormalities (submucosal fibroids, intramural fibroids greater than 3 cm in diameter, large subserosal fibroids, endometrial polyps);
2. laboratory abnormalities (follicle-stimulating hormone level higher than 40 iu/l, adverse endometrial histology)
3. hysteroscopic abnormalities (submucosal fibroids, endometrial polyps),
4. incidental adnexal abnormality on ultrasound,
5. severe intermenstrual bleeding, severe dysmenorrhoea, severe premenstrual pain, chronic pelvic pain,
6. medical contraindications to either study treatment,
7. previous endometrial ablation or resection,
8. uninvestigated postcoital bleeding
9. untreated abnormal cervical cytology.
10. pregnancy; lactation; occurrence of <3 menstrual cycles following childbirth, abortion or lactation;
11. current use of an intrauterine device; hypersensitivity to any of the study drug ingredients and known or suspected malignant or premalignant disease.
12. systemic diseases like hypertension, diabetes, thyroid diseases or coronary artery diseases; and history of previous medication for menorrhagia
13. using anticoagulant drugs

Ages: 40 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women who were admitted to our outpatient clinic with heavy menstrual bleeding aged 40 to 50 years old and treated with e2v/dng, lng-ıud or oral micronized progesterone.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: cihan kaya, Study Director — Bakırkoy Dr. Sadi Konuk Training and Research Hospital
Locations (1):
- Bakirkoy Dr. Sadi Konuk Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Estradiol Valerate: Women who were treated with Estradiol valerate for Heavy Menstrual Bleeding for 3 months.
- LNG-IUD: Women who were treated with Levonorgestrel Intrauterine Device (LNG-IUD) for Heavy Menstrual Bleeding for 4 years.
- Micronized Progesterone: Women who were treated with Micronized Progesterone for Heavy Menstrual Bleeding for 3 months.
Period: Overall Study
Arm/Group | Estradiol Valerate | LNG-IUD | Micronized Progesterone
Started | 37 | 33 | 34
Completed | 37 | 33 | 34
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- LNG-IUD: Women who were treated with Levonorgestrel Intrauterine Device LNG-IUD for Heavy Menstrual Bleeding for 4 years.
- Total: Total of all reporting groups
Arm/Group | Estradiol Valerate | LNG-IUD | Micronized Progesterone | Total
Number analyzed (Participants) | 37 | 33 | 34 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.7 (4.7) | 45 (4.6) | 45.4 (4.7) | 45 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 33 | 34 | 104
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Hot Flush Frequency Total Score (HFRS) Change
Description: Hot flush rating scale (HFRS) is a 5 items subjective tool. The first and second items of this scale are for Hot Flush Frequency Score. Women were asked to provide ratings of the frequency of hot flushes and night sweats in the first and second items. The number of the frequency in the first and second item is summed and this score is the total hot flush frequency score. The minimum Hot Flush Frequency Score is 0 and there is no maximum score to provide. However, the higher scores represent worse outcome. In this study, the Hot Flush Frequency Score is measured and recorded at initial of the treatment and six months of treatment. The change between the initial and six months score is our first primer outcome.
Time Frame: change from initial hot flush frequency score at 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Estradiol Valerate | LNG-IUD | Micronized Progesterone
Number analyzed (Participants) | 37 | 33 | 34
score on a scale | 9.3 (26.4) | 8.8 (20.5) | 12.7 (30.3)

2. Primary Outcome: Total Menopause Rating Scale (MRS) Score Change
Description: Menopause Rating Scale (MRS) is a questionnaire that assesses the presence and intensity of 11 menopausal symptoms. These are grouped into three subscales: the somatic subscale, the psychological subscale and the urogenital subscale. Each of the 11 items can be rated by the participant from 0 (not present) to 4 (very severe). The scores obtained for each individual item are summed to provide the corresponding total subscale score. The sum of subscales scores provide the total MRS score. Higher scores are indicative of more severe symptoms. Minimum total MRS score is 0 and maximum total MRS score is 44.
Time Frame: change from initial menopause rating scale score at 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Estradiol Valerate | LNG-IUD | Micronized Progesterone
Number analyzed (Participants) | 37 | 33 | 34
score on a scale | -0.4 (6.5) | -2.5 (7.4) | -1.4 (4.7)

3. Secondary Outcome: Menopause Multi-Attribute Score Change on Menopause Multi-Attribute Scale.
Description: This is measured by menorrhagia multi-attribute scale; which is designed to measure the effect of menorrhagia on six domains of daily life (practical difficulties, social life, psychological health, physical health, work and daily routine, and family life and relationships). Scores range from 0 (severely affected) to 100 (not affected). Higher scores represent a better outcome.
Time Frame: change from initial menopause multi-attribute score at 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Estradiol Valerate | LNG-IUD | Micronized Progesterone
Number analyzed (Participants) | 37 | 33 | 34
score on a scale | 25.2 (31.1) | 31.0 (26.7) | 22.8 (26.7)

4. Secondary Outcome: Pictorial Bleeding Assessment Score Change
Description: The pictorial blood assessment chart (PBAC) consists of a series of diagrams representing lightly, moderately, and heavily soiled towels and tampons. The numbers at the top of the chart represent the day of menstruation. The women are instructed to insert a mark in the appropriate box at the time each towel and/or tampon is discarded. After completion, the woman returns the chart during her next appointment to the clinic. The chart is scored using the scoring system. A baseline score is established and then at six months of treatment, the score is assessed again. Change from the initial score at 6 months of treatment is recorded as a secondary outcome. Decreasing values are considered to be a better outcome.
Time Frame: change from initial Pictorial bleeding assessment score at 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Estradiol Valerate | LNG-IUD | Micronized Progesterone
Number analyzed (Participants) | 37 | 33 | 34
score on a scale | -113 (61.6) | -120.7 (51.2) | -112.5 (54.8)

5. Secondary Outcome: Hemoglobin Value Change
Description: Blood sample analysis for hemoglobin values is performed before the treatment and at six months of treatment.
Time Frame: change from initial hemoglobin values at 6 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Estradiol Valerate | LNG-IUD | Micronized Progesterone
Number analyzed (Participants) | 37 | 33 | 34
mg/dL | 0.5 (1.2) | 0.09 (1.4) | 0.03 (1.4)

ADVERSE EVENTS:
Time Frame: 12 months
Description: There was no adverse event.
Arm/Group | Estradiol Valerate | LNG-IUD | Micronized Progesterone
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/33 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/33 | 0/34
Other Adverse Events (participants affected / at risk) | 0/37 | 0/33 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT03368898/Prot_SAP_000.pdf